CLINICAL TRIAL: NCT02787083
Title: A Pilot Study of the Effects of Mirabegron on Symptoms in Patients With Interstitial Cystitis
Acronym: MirabegronIC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Philadelphia Urosurgical Associates (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Principal Investigator, Kristene Whitmore, MD, Philadelphia Urosurgical Associates
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MYRB-15G02
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Cystitis, Interstitial
Keywords: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirabegron (Experimental): These patients will receive mirabegron 50mg tablets daily for 12 weeks.
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator): These patients will receive placebo tablets daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron
  Other Names: Myrbetriq
  Arms: Mirabegron
Drug: Placebo
  Arms: Placebo

SUMMARY:
Bladder pain syndrome/interstitial cystitis (BPS/IC) is a difficult disease to both diagnose and treat. It is defined as an unpleasant sensation (pain, pressure, or discomfort) perceived to be related to the urinary bladder and associated with lower urinary tract symptoms for at least 6 weeks duration, in the absence of infection or other identifiable causes. Pain is the universal symptom, but many also experience symptoms of overactive bladder, possibly directly related to the mechanism of pain. Treating pain may influence the symptom of urgency, if the urge arises from a need to alleviate pain. In some patients whose pain improves with treatment, troubling overactive bladder symptoms still remain. Beta-3 adrenergic agonists have been found to decrease signaling of C-fibers in animal models. So, the investigators hypothesize that mirabegron, which is FDA-approved for treatment of overactive bladder, would also improve symptoms in patients with BPS/IC. As a selective beta-3 agonist, mirabegron acts on the beta-3 receptors found in the bladder which mediate relaxation of the detrusor muscle. It has been shown to significantly decrease the number or micturition episodes, urgency episodes, and increased mean volume of urine voided per micturition. It also has a favorable tolerability profile.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be diagnosed with BPS/IC with a minimum O'Leary-Sant score of 8 on the ICSI, as well as 8 on the ICPI. Participants should be stable on their regimen (no increase or change in medications, behavioral treatments or physical therapy in previous 4 weeks prior to starting the study) and be willing to remain on this regimen during the duration of the study.

   1. Participant must be stable on current IC/BPS regimen.
   2. Participant must have subjective complaints of

   i. urinary urgency, relieved with voiding or ii. urinary frequency; ≥ 8 voids per day iii. pelvic pain, pressure, hypersensitivity or discomfort
2. Gender of subjects: Participants in this study will be female. Pregnant women and breastfeeding women will be excluded due to unknown risk of study medication on pregnancy and fetus or nursing infants.
3. Age of subjects: Age of participants will range from 18 to 95 years.
4. Racial and ethnic origin: There are no enrollment restrictions based upon race or ethnic origin. The racial and ethnic distribution of participants is entirely based on the population of patients at the study site.
5. Other inclusion criteria:

   1. Participant must give written informed consent to participate in the study
   2. Participant must be able to make decisions for herself
   3. Participant must have a negative urine dip within 7 days prior to start of the study
   4. Female participants who are of childbearing age and sexually active with men must agree to use a medically acceptable method of contraception throughout the study period, and for 7 days after the study period. Medically acceptable methods of contraception include abstinence, oral contraceptive pills, hormonal contraceptive patches, diaphragm with or without spermicide, IUD, condoms, depot medroxyprogesterone acetate, subdermal progestin implants, vasectomized partner, or status post surgical sterilization.

Exclusion Criteria:

To participate in the study subjects must not meet any of the following criteria:

1. Participant is currently pregnant or breastfeeding
2. Participant has a positive urinary pregnancy test at the time of screening
3. Participant is currently or has been on antibiotic therapy with the last 7 days prior to the start of the study
4. Participant is an employee of Astellas, or any other pharmaceutical company or the Pelvic and Sexual Health Institute
5. Participant is currently in another pharmaceutical trial
6. Participant has used anticholinergic medications, tamsulosin or opioid narcarotic medication within the last 30 days prior to the study or during the study period. Participants will be able to use rescue medications for BPS/IC symptom flares including non-opioid narcotics, non-steroidal anti-inflammatory agents, pyridium and uribel.
7. Participant has had bladder hydrodistention or bladder instillations within the last 4 weeks. Participants may have bladder instillations during the study period if necessary for rescue from symptom flares.
8. Participant has used or currently using CYP2D6 substrates, such as thioridazine, flecainide, propafenone, within the last 7 days prior to the study or during study period
9. Participant has used warfarin or digoxin within the last 7 days prior to the study or during the study period
10. Participant has used cyclosporine within the 7 days prior to the study or during the study period
11. Participant has an active S3 nerve stimulator implanted or has had PTNS within 6 months prior to starting the study
12. Participant has not had intravesical botulinum toxin injection in 6 months prior to starting the study
13. Participant has grade III or IV pelvic organ prolapse
14. Participant has been diagnosed with a urinary tract infection within the last 4 weeks prior to starting the study
15. Participant has history of bladder cancer
16. Participant is currently an alcohol or substance abuser, or is a chronic opioid user
17. Participant has history of renal failure (GFR <30) or liver failure (CHILD score B or C)
18. Participant has urinary retention defined as greater than 150cc post-void residual as diagnosed by catheterization, bladder ultrasound scan or urodynamic testing within the last 14 days.
19. Participant has history of severe uncontrolled blood pressure (defines as systolic greater than or equal to 180mm Hg and/or diastolic blood pressure greater than or equal to 110 mm Hg)
20. Participant has a neurological disease including, but not limited to, multiple sclerosis, Parkinson's disease, Alzheimer's disease, spinal cord injury, brain injury, stroke or dementia
21. Participant has urinary frequency of less than 8 times/day
22. Participant has bladder or lower ureteral calculi
23. Participant has active genital herpes
24. Participant has urethral diverticulum
25. Participant has chemical cystitis
26. Participant has radiation or tuberculosis cystitis
27. Participant has known hypersensitivity to mirabegron or any of the inactive ingredients in the supplied form of mirabegron

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08; Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristene E Whitmore, MD, Study Director — Philadelphia Urosurgical Associates
Locations (1):
- Philadelphia Urosurgical Associates, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirabegron: These patients will receive mirabegron 50mg tablets daily for 12 weeks.
  Mirabegron
- Placebo: These patients will receive placebo tablets daily for 12 weeks.
  Placebo
Period: Overall Study
Arm/Group | Mirabegron | Placebo
Started | 4 | 5
Completed | 1 | 3
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9
Systolic [Mean (Full Range); unit: MMHg] | 145 [110 to 180] | 145 [110 to 180] | 145 [110 to 180]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Interstitial Cystitis Symptom Improvement
Description: Evaluate urinary urgency, frequency and pain via validated O'Leary Sant questionnaire
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 1 | 3
Participants | 1 | 3

2. Secondary Outcome: Number of Participants With Improvement in Incontinence Episodes
Description: Evaluate incontinence episodes via bladder diary and UDI-6 questionnaire
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 1 | 3
Participants | 1 | 3

3. Secondary Outcome: Impact on Quality of Life
Description: Evaluate impact on quality of life from bladder, bowel and vaginal/pelvic symptoms via PFIQ-7 questionnaire
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Patient Satisfaction
Description: evaluate participant satisfaction with treatment/placebo via Global response assessment form
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Sexual Function
Description: Evaluate changes in sexual function via FSFI questionnaire
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Side Effects of Medication
Description: Will assess if participants have side effects of medication via office visits
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse event happened in the beginning of the study within a 3 month period.
Description: The participants were all healthy adults
Arm/Group | Mirabegron | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 1/4 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=4) | Placebo (N=5)
Headache (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT02787083/Prot_SAP_ICF_000.pdf